CLINICAL TRIAL: NCT06720519
Title: Multiparametric Molecular Panel Evaluation "QIAstatDxMeningitis/Encephalitis" for Diagnosis of Infections of the Central Nervosous System
Brief Title: Molecular Panel Evaluation for Diagnosis of Infections of the Central Nervosous System
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: QIA-ME; 2024/67 QIAMA (Other Grant/Funding Number: QIAGEN STAT-Dx Life S.L)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Infections Nervous System
Keywords: Central nervous system infections; Bacterial Infection; Viral Infection; Meningitis; Encephalitis
MeSH Terms: conditions — Central Nervous System Infections; Bacterial Infections; Virus Diseases; Meningitis; Encephalitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Positive Samples: Positive samples for viruses or bacteria typical of meningitis/encephalitis
  Interventions: Diagnostic Test: QIAstat-Dx®Meningitis/Encephalite Panel

INTERVENTIONS:
Diagnostic Test: QIAstat-Dx®Meningitis/Encephalite Panel — The analytical sensitivity of the test is assessed by comparing the results obtained with those known from routine diagnostic tests.
  For viruses only, the semi-quantitative value of Ct is also evaluated with the viral load provided by qPCR.

SUMMARY:
Infections involving the central nervous system (CNS), such as meningitis/encephalitis (ME), are serious clinical conditions associated with high morbidity and mortality rates, as well as significant long-term consequences. ME can be caused by a wide variety of pathogenic agents. Clinical symptoms may vary and it has been shown that early identification of the pathogens causing ME allows for timely and appropriate treatment, thus reducing permanent neurological damage. The multiparameter panel "QIAstat-Dx®Meningitis/Encephalitis" can detect in one hour on a sample of 15 bacterial, viral and fungal pathogens. In the diagnostic routine, Real-time PCR takes an average of 3 hours and culture examination 2 days. In addition, compared to other comparable rapid molecular systems, the "QIAstat-Dx" platform has the ability to generate a cycle-related threshold value (Ct) for the targets detected. This value may have a correlation with the viral load and thus provide in a short time not only the result of positivity, but also an indication of the amount of virus present. Other commercially available multiparameter molecular tests provide only qualitative data.

DETAILED DESCRIPTION:
The study is on biological samples of cerebrospinal fluid, positive for viruses or bacteria of interest, retrospective, monocentric, non-pharmacological.

For each sample included in the study (170 total samples), the molecular/culture test result, provided by the normal diagnostic process at the Microbiology Unit, is available for comparison with those obtained with the multiparameter panel QIAstat-Dx® Meningitis/Encephalitis (ME) and QIAstat-Dx 1.0 analyzer.

The aim of the study is:

1. To evaluate the analytical sensitivity of the test by identifying positive samples for bacteria (culture comparison) and positive samples for viruses (qPCR comparison).
2. Compare the value of Ct obtained with the number of viral copies per ml of cerebrospinal fluid obtained by qPCR.

ELIGIBILITY:
Inclusion Criteria:

* 170 samples of CSF positive for virus and/or bacteria;
* Samples stored at -80°C, less than 5 years;
* Samples with a volume of at least 800μL.

Exclusion Criteria:

* Samples of a different matrix than CSF;
* Samples stored at room temperature;
* Samples for which diagnostic test results are not available;
* Samples with a volume of less than 800μL;
* Samples already thawed and refrozen.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Virus or bacterial positive samples from cerebrospinal fluid.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The analytical sensitivity of the multiparameter panel | 6 months
  The analytical sensitivity of the test is assessed by comparing the results obtained with those known from routine diagnostic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Gabrielli, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Penata A, Mesa S, Leal A, Castano T, Bustamante J, Sigifredo O. Molecular diagnosis of meningitis and meningoencephalitis with an automated real-time multiplex polymerase chain reaction in a tertiary reference complex in Medellin, Colombia. Rev Inst Med Trop Sao Paulo. 2020 Oct 9;62:e77. doi: 10.1590/S1678-9946202062077. eCollection 2020. PMID 33053146
- [Background] Shin SY, Kwon KC, Park JW, Kim JM, Shin SY, Koo SH. Evaluation of the Seeplex(R) Meningitis ACE Detection kit for the detection of 12 common bacterial and viral pathogens of acute meningitis. Ann Lab Med. 2012 Jan;32(1):44-9. doi: 10.3343/alm.2012.32.1.44. Epub 2011 Dec 20. PMID 22259778
- [Background] Messacar K, Breazeale G, Robinson CC, Dominguez SR. Potential clinical impact of the film array meningitis encephalitis panel in children with suspected central nervous system infections. Diagn Microbiol Infect Dis. 2016 Sep;86(1):118-20. doi: 10.1016/j.diagmicrobio.2016.05.020. Epub 2016 Jun 2. PMID 27342782
- [Background] Leber AL, Everhart K, Balada-Llasat JM, Cullison J, Daly J, Holt S, Lephart P, Salimnia H, Schreckenberger PC, DesJarlais S, Reed SL, Chapin KC, LeBlanc L, Johnson JK, Soliven NL, Carroll KC, Miller JA, Dien Bard J, Mestas J, Bankowski M, Enomoto T, Hemmert AC, Bourzac KM. Multicenter Evaluation of BioFire FilmArray Meningitis/Encephalitis Panel for Detection of Bacteria, Viruses, and Yeast in Cerebrospinal Fluid Specimens. J Clin Microbiol. 2016 Sep;54(9):2251-61. doi: 10.1128/JCM.00730-16. Epub 2016 Jun 22. PMID 27335149
- [Background] de Crom SC, Obihara CC, van Loon AM, Argilagos-Alvarez AA, Peeters MF, van Furth AM, Rossen JW. Detection of enterovirus RNA in cerebrospinal fluid: comparison of two molecular assays. J Virol Methods. 2012 Jan;179(1):104-7. doi: 10.1016/j.jviromet.2011.10.007. Epub 2011 Oct 15. PMID 22024398
- See also: Emergency management in bacterial meningitis and sepsis: application of real time-polymerase chain reaction and FilmArray technology performed directly on cerebrospinal fluid and blood samples Authors Loria Bianchi — https://www.pagepressjournals.org/mm/article/view/5084
- See also: Role of computed tomography before lumbar puncture: a survey of clinical practice — https://pmc.ncbi.nlm.nih.gov/articles/PMC2117486/